CLINICAL TRIAL: NCT06918119
Title: Characterization of Transcutaneous Spinal Cord Stimulation for Enabling Reflex Motor Evoked Responses in Children and Youth With Spina Bifida
Brief Title: Transcutaneous Spinal Stimulation for Children and Youth With Spina Bifida
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 24-006063
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Myelomeningocele; Spina Bifida
MeSH Terms: conditions — Meningomyelocele; Spinal Dysraphism | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Functional motor training with transcutaneous spinal cord stimulation (Experimental): Transcutaneous spinal cord stimulation will be delivered to the skin over the lower thoracic and lumbar spine region using adhesive electrodes for ages 5-11 for one multi-hour visit. The effects of stimulation will be recorded via electrophysiological and biomechanical metrics described within the outcomes measures.
  Interventions: Device: Transcutaneous stimulation
- Extended functional motor training with transcutaneous spinal cord stimulation (Experimental): An extended functional training arm for a subset of 10 subjects, ages 12-18, in which they will receive up to twelve multi-hour sessions of a therapeutic neuromuscular strengthening intervention within a 6 week period.
  Interventions: Device: Transcutaneous stimulation

INTERVENTIONS:
Device: Transcutaneous stimulation — DS8R (Digitimer LLC) for transcutaneous neurostimulation.

SUMMARY:
A study to use transcutaneous spinal cord stimulation to characterize sensorimotor deficits in a pediatric population of individuals with spina bifida.

DETAILED DESCRIPTION:
The study's goals involve understanding how transcutaneous stimulation affects motor deficits across three dimensions; weakness, coordination, and spasticity. This will be investigated by an electrophysiological characterization lower-extremity deficits, using TS to interrogate neuromotor topography and connectivity of the spinal cord to specific muscles. These evaluations will enable a unique patient-specific understanding of the electrophysiological mechanisms underlying motor deficits. Furthermore, these evaluations will assess the therapeutic potential of a novel closed-loop TS plasticity induction protocol to strengthen weakened muscles in a pediatric SB population.

ELIGIBILITY:
Inclusion Criteria

* Congenital diagnosis of myelomeningocele (MMC)
* Able to follow verbal commands or instructions.
* If female and able to become pregnant, must be willing to use medically-acceptable method of contraception during study participation.

Exclusion Criteria

* Severe cognitive deficits demonstrating inability to communicate needs
* Gaping, weeping, or unhealed open wounds at the site of electrode placement
* Unhealed fractures on load bearing bones
* History of osteoporosis
* History of implanted electronic devices at the stimulation location(e.g. deep brain stimulator, cardiac pacemaker, diaphragmatic pacer, baclofen pumps, insulin pumps, etc.)
* Pregnancy
* Epilepsy
* History of seizure
* Ongoing infections (currently being treated or are symptomatic)
* Any illness or condition which, based on the research team's assessment, will compromise the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Manual muscle testing (MMT) | 1 to 12 visits (up to 6 weeks)
  Measuring muscle strength and function using the Daniels and Worthingham's Muscle Grading Scale. A physical therapist will use a 5-point scale to manually test the 5 lower extremity muscles on each side, with 0 being no visible or palpable contraction, up to 5 being full range of motion against gravity with maximal resistance. The maximum total score would be 50.
Spasticity (1) | 1 to 12 visits (up to 6 weeks)
  Change in measurement of leg muscle tone utilizing the Modified Ashworth Scale (MAS). A physical therapist will use a 5-point scale to assess resistance of major muscles during passive range of motion, with a lower score for a muscle indicating less tone. MAS for 4 muscle groups in each leg will be reported.
Spasticity (2) | 1 to 12 visits (up to 6 weeks)
  Change in measurements of leg muscle tone utilizing Wartenberg's pendulum test, with the first swing angle (FSA) degrees as the primary outcome. Fewer degrees on swing angle indicating greater spasticity.
Gait | 1 to 12 visits (up to 6 weeks)
  Gait speed will be quantified in m/sec utilizing a motion capture system, with faster gait speed indicating less impairment.
Coordination | 1 to 12 visits (up to 6 weeks)
  Coordination will be reported with the Selective Control Assessment of the Lower Extremity (SCALE) total limb score for both right and left leg. Total score for each limb is 10, with a higher score indicating coordination closer to optimal.

SECONDARY OUTCOMES:
Electromyography (EMG) | 1 to 12 visits (up to 6 weeks)
  TS-evoked motor potential (MEP) amplitude, in millivolts, will be reported for major lower limbs muscles. An increase in MEP amplitude is indicative of greater muscle activation, closer to optimal function.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Zhao, Ph.D., Principal Investigator — Mayo Clinic; Joline Brandenburg, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.